CLINICAL TRIAL: NCT04865107
Title: Cellular Immuno-Therapy for COVID-19 ARDS Randomized Clinical Trial
Acronym: CIRCA-19 RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIRCA-19 RCT
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Covid19; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized (2:1) placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSCs Arm (Experimental): 3 daily doses of up to 90-million cells/unit dose (cumulative dose of up to 270 million UC-MSCs)
  Interventions: Biological: UC-MSCs
- Placebo Arm (Placebo Comparator): 3 daily doses of up to 90-million cells/unit dose (cumulative dose of up to 270 million UC-MSCs)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UC-MSCs — 3 daily doses of up to 90-million cells/unit dose (cumulative dose of up to 270 million UC-MSCs)
  Arms: MSCs Arm
Biological: Placebo — PlasmaLyte A and 5% Human Albumin
  Arms: Placebo Arm

SUMMARY:
This is a Phase 2 multicenter randomized (2:1), placebo-controlled trial to evaluate early signs of efficacy of allogeneic, umbilical cord-derived (UC) mesenchymal stromal cells (MSCs) in patients with COVID-19 and Acute Respiratory Distress Syndrome (ARDS).

Randomized participants (N=54) will receive 3 daily doses of up to 90-million cells/unit dose (cumulative dose of up to 270 million UC-MSCs) or blinded placebo. The MSC product will be provided as 2.5 million cells/ml suspended in PlasmaLyte A containing 5% Human Albumin. The appearance-matched placebo product contains the same excipients, PlasmaLyte A and 5% Human Albumin, as the UC-MSCs.

ELIGIBILITY:
Inclusion Criteria:

* Age of ≥18 years
* Laboratory-confirmed SARS-CoV-2 infection during the current admission
* On invasive, non-invasive mechanical ventilation (NIV) (PEEP ≥5 cmH20) or high-flow nasal canula (HFNC) oxygen therapy (minimum total flow rate of 40 lpm)
* ARDS (onset <96h) as per the international consensus definition (P/F ratio < 300 with PEEP ≥5cm H20 or on HFNC), not due primarily to cardiac causes.

Exclusion Criteria:

* No consent/inability to obtain consent
* Rockwood Clinical Frailty Score > 4
* Moribund patient not expected to survive 24 hours
* Any other irreversible disease or condition for which 6-month mortality is estimated to be greater than 50%
* Currently receiving extracorporeal life support
* Pregnant or lactating
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Moderate to severe chronic liver disease (Childs-Pugh Score > 12)
* Severe chronic respiratory disease with a baseline PaCO2 > 50 mm Hg or the use of home oxygen
* Documented deep venous thrombosis or pulmonary embolism within the preceding 3 months
* Inability/contra-indications to receiving local standard of care thromboprophylaxis
* Chronic immunosuppression (any chronic immunotherapy including daily oral steroid use >6months)
* Known HIV, Hep B/C positive, or active tuberculosis
* Multisystem shock (SOFA score change from baseline of >2 in >2 systems)
* Patient, surrogate, or physician not committed to full support including intubation (exception: a patient will not be excluded if he/she would receive all supportive care except for attempts at resuscitation from cardiac arrest)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Number of days free of oxygen by NIV/HFNC or mechanical ventilation at Day 28 | Day 28

SECONDARY OUTCOMES:
Biomarkers of systemic inflammatory response | Change from Baseline to 24 hours after each MSC infusion
  Interleukin levels change from Baseline to 24 hours after each MSC infusion
Biomarkers of endothelial function | Change from Baseline to 24 hours after each MSC infusion
  Angiopoietin levels change from Baseline to 24 hours after each MSC infusion
ICU mortality | Day 28
  Number of deaths at day 28

OTHER OUTCOMES:
Safety events (SAEs, AEs) | At time of infusion until one year post-infusion
  allergic reactions, infusion related reactions, and venous and arterial thrombotic events

CONTACTS AND LOCATIONS:
Overall Officials: Duncan J Stewart, MD, Principal Investigator — The Ottawa Hospital
Locations (4):
- Canada (4):
  - Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No